CLINICAL TRIAL: NCT06884280
Title: Proactive High Dose Versus Low-dose Reactive Intravenous or Oral Iron in People on Peritoneal Dialysis (PALaDIN) - an Open-label, Feasibility Randomised Study
Brief Title: Comparing High and Low Dose Iron Treatments for People on Peritoneal Dialysis: The PALaDIN Study
Acronym: PALaDIN
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Collaborators: Pharmacosmos Therapeutics, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R4171
Record Dates: First submitted 2025-02-10; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-02

CONDITIONS: Peritoneal Dialysis; Anaemia; Iron Deficiency, Anaemia
MeSH Terms: conditions — Anemia; Anemia, Iron-Deficiency | interventions — iron isomaltoside 1000; ferric derisomaltose; ferrous sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oral (Active Comparator): Ferrous Sulphate 200mg once daily (oral)
  Interventions: Drug: Ferrous Sulfate
- Reactive Intravenous (Experimental): IV Monofer up to every 3 months. Administered if ferritin <100 ug/L and TSAT <20%
  Interventions: Drug: Monofer (iron isomaltoside 1000)
- Proactive Intravenous (Experimental): IV Monofer up to every 3 months. Administered if ferritin <700 ug/L and TSAT <40%
  Interventions: Drug: Monofer (iron isomaltoside 1000)

INTERVENTIONS:
Drug: Monofer (iron isomaltoside 1000) — Intravenous iron infusion, administered in this study up to every 3 months. Dosage determined by haemoglobin and weight.
  Other Names: Ferric derisomaltose
  Arms: Proactive Intravenous; Reactive Intravenous
Drug: Ferrous Sulfate — Oral iron tablet taken once daily for duration of study.
  Arms: Oral

SUMMARY:
Chronic kidney disease affects a significant portion of the UK population, with approximately 3.5 million adults diagnosed. At its most severe stage, end-stage kidney disease, individuals require frequent dialysis treatment. One form of dialysis, known as peritoneal dialysis, involves introducing and removing fluid from the abdominal cavity to help filter out toxins from the body.

The kidneys are involved in various hormonal processes, including those responsible for producing red blood cells, making anaemia a common consequence of kidney failure. When designing a clinical trial to evaluate the effectiveness of any treatment, it is essential to determine the number of suitable and willing participants, as well as those who can complete all required tests and measurements. Identifying the most appropriate measurement to assess the impact of intravenous iron (iron injected directly into veins) is crucial to ensure that any observed changes are meaningful to people with CKD and their carers. To address these considerations, the investigators will conduct a pilot feasibility trial.

In this trial, individuals with kidney disease undergoing peritoneal dialysis will be randomly assigned to receive either high-dose or low-dose intravenous iron, or oral iron therapy. Over twelve months, the investigators will monitor their anaemia response, symptoms of kidney disease, quality of life, physical performance (such as the ability to walk for six minutes), and cognitive function. Additionally, the investigators will assess the impact of each intervention on the frequency of blood transfusions, whether those on oral iron require intravenous iron, and any changes in the dosage of erythropoietin-stimulating agents (drugs that increase blood production).

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged ≥18 years.
* Able to give informed consent
* Serum ferritin <700ug/L
* Transferrin saturation level <40%
* No intravenous iron for last 4 weeks before randomisation (patients may be pre-identified and included after 4-week washout period)
* Received maintenance peritoneal dialysis therapy for at least 4 weeks
* Expected to remain on peritoneal dialysis therapy for duration of study

Exclusion Criteria:

* Inadequate dialysis deemed by responsible clinician
* Probability of need for transfusion within 1 week of enrolment
* Anticipated major surgery that the responsible clinician feels will impact response to treatment
* Haemochromatosis / haemosiderosis or ALT >x3 normal
* Are deemed to be most suited to best-supportive or end-of-life care at time of screening
* Women of childbearing potential not using effective means of contraception
* Have been involved in another medicinal study (CTIMP) within past 4 weeks
* Known allergy or adverse reaction to oral or intravenous iron preparations
* CRP >50, TSATs >40%, SF >700 at time of recruitment
* Active infection, HIV, active Hep B or C
* Are unable or unwilling to consent to or complete the study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Eligibility to consent rate (%) | From enrollment to the end of treatment at 12 months
  This refers to the proportion of participants who are eligible for the study and who provide informed consent to participate.
  Measuring Eligibility to Consent Eligibility-to-Consent Rate: (Number of eligible participants who consented / Total number of eligible participants) × 100% A low eligibility-to-consent ratio may suggest challenges in participant engagement, while a high ratio indicates good participant willingness to take part.
Recruitment rate (%) | From enrollment to the end of treatment at 12 months
  The recruitment rate refers to the speed at which participants are enrolled into a study over a given time period.
  Measuring Recruitment Rate Recruitment Rate: (Number of participants enrolled / Time period, e.g., per month)
  For multi-site studies, it can be adjusted per site:
  Recruitment Rate per Site: (Total participants enrolled / Number of sites × Time period) A high recruitment rate suggests effective recruitment strategies, while a low rate may highlight recruitment barriers.
Participant retention to 12 month follow-up (%) | From enrollment to the end of treatment at 12 months
  Participant retention refers to the proportion of participants who remain in the study and complete follow-up assessments over time.
  Measuring Retention Retention Rate at Follow-Up: (Number of participants completing follow-up assessments / Total participants enrolled) × 100% A high retention rate reflects good participant engagement, while a low rate may suggest challenges such as participant burden or study fatigue.
Completion of clinical outcomes at follow-up and patterns of missing data for the study measures (%) | From enrollment to the end of treatment at 12 months
  This refers to the proportion of participants who complete the clinical outcomes measures at follow-up.
  Measuring Completion of Clinical Outcomes Completion Rate of Clinical Outcomes: (Number of participants with complete clinical outcome data / Total participants expected at follow-up) × 100% This measures how well the study is able to collect necessary data, with a high completion rate indicating effective data collection processes.
Completion of patient symptom questionnaires throughout the study (%) | From enrollment to the end of treatment at 12 months
  This refers to the proportion of scheduled symptom questionnaires that participants complete during the study. It is an important measure of participant engagement and the completeness of patient-reported outcome data.
  Measuring Completion of Patient Symptom Questionnaires Questionnaire Completion Rate: (Number of completed questionnaires / Total number of expected questionnaires) × 100% A high completion rate indicates good participant involvement and reliable data, while a low rate may suggest that the questionnaires are burdensome, inconvenient, or not seen as valuable by participants.
Treatment adherence (%) | From enrollment to the end of treatment at 12 months
  Treatment adherence refers to how well participants follow the prescribed treatment regimen, whether it is medication, lifestyle changes, or other interventions.
  Measuring Adherence Adherence Rate: (Number of prescribed doses/sessions completed / Total prescribed doses/sessions) × 100% A high adherence rate indicates good compliance, while a low rate may indicate barriers such as treatment side effects, participant preference, or complexity of the regimen.
Treatment fidelty (%) | From enrollment to the end of treatment at 12 months
  Treatment fidelity refers to the degree to which the intervention is delivered as per the study protocol, ensuring consistency across all participants and study sites.
  Measuring Fidelity Fidelity Rate: (Number of intervention components delivered as intended / Total expected intervention components) × 100% A high fidelity rate suggests that the intervention is being delivered consistently as intended, while a low rate may indicate deviations in protocol delivery.
Treatment acceptability (%) | From enrollment to the end of treatment at 12 months
  Treatment acceptability refers to how acceptable participants or healthcare providers find the study intervention, including factors such as ease of use, side effects, and perceived effectiveness.
  Measuring Acceptability Acceptability Rate: (Number of participants rating treatment as acceptable / Total participants assessed) × 100% Acceptability is often measured through surveys or questionnaires, and a high rate indicates that participants find the treatment tolerable and beneficial. Low acceptability may highlight barriers such as side effects or perceived inefficacy.

SECONDARY OUTCOMES:
Adverse and serious adverse events | From enrollment to the end of treatment at 12 months
  Adverse Events (AEs) An adverse event (AE) is any unwanted or harmful medical occurrence in a participant receiving a study intervention, regardless of whether it is directly related to the intervention. This includes symptoms, abnormal lab findings, or worsening of an existing condition.
  Measuring AEs Incidence Rate: (Number of participants experiencing at least one AE / Total participants enrolled) × 100% AE Frequency: Total number of AEs / Total participants enrolled Severity Grading: Often classified as mild, moderate, or severe based on clinical criteria (e.g., CTCAE grading system).
Mortality and Major Adverse Cardiovascular Events (MACE) | From enrollment to the end of treatment at 12 months
  Mortality and Major Adverse Cardiovascular Events (MACE) Mortality refers to the number of deaths occurring in the study population. Major Adverse Cardiovascular Events (MACE) typically include cardiovascular death, non-fatal myocardial infarction, non-fatal stroke, and heart failure hospitalisation.
  Measuring Mortality and MACE Mortality Rate: (Number of deaths / Total participants enrolled) × 100% MACE Incidence Rate: (Number of participants experiencing at least one MACE / Total participants enrolled) × 100% Event-Specific Rates: Tracking occurrences of cardiovascular death, myocardial infarction, stroke, and heart failure admissions separately.
Hospital Admissions | From enrollment to the end of treatment at 12 months
  This includes any unplanned or planned hospitalisations occurring during the study period. It is a key measure of disease burden and healthcare utilisation.
  Measuring Hospital Admissions Hospital Admission Rate: (Number of participants admitted to hospital / Total participants enrolled) × 100% Admission Frequency: Total number of hospital admissions / Total participants enrolled Length of Stay: Average number of days spent in hospital per admission
Drug Reactions | From enrollment to the end of treatment at 12 months
  This includes any adverse reactions or side effects experienced by participants due to study medication. Reactions can range from mild to severe, including life-threatening anaphylaxis or organ toxicity.
  Measuring Drug Reactions Incidence Rate: (Number of participants experiencing at least one drug reaction / Total participants receiving the drug) × 100% Severity Grading: Categorising reactions as mild, moderate, severe, or life-threatening Causality Assessment: Evaluating whether the reaction is likely related to the study drug
Infections and Peritoneal Dialysis Peritonitis | From enrollment to the end of treatment at 12 months
  This includes any infections occurring during the study, with a specific focus on peritoneal dialysis (PD) peritonitis, a serious complication in PD patients.
  Measuring Infections and PD Peritonitis Infection Rate: (Number of participants experiencing at least one infection / Total participants enrolled) × 100% PD Peritonitis Rate: Number of peritonitis episodes / Total PD patient-months Pathogen Identification: Categorising infections based on microbiological findings (e.g., Gram-positive, Gram-negative, fungal) Antibiotic Response Rate: (Number of resolved infections with first-line antibiotics / Total treated infections) × 100%
Quality of life (KDQoL-SF) | From enrollment to the end of treatment at 12 months
  Quality of life (QoL) refers to participants' overall well-being, encompassing physical, emotional, and social aspects of life. It is typically measured using validated tools or disease-specific instruments (KDQoL-SF)
  Measuring Quality of Life QoL Score: (Sum of individual item scores / Total possible score) × 100% Higher scores indicate better quality of life, while lower scores suggest poorer well-being.
Symptom burden (IPOS-Renal, PROMIS Global Health Instrument) | From enrollment to the end of treatment at 12 months
  Symptom burden refers to the overall impact of symptoms on a participant's daily life, including severity, frequency, and the level of distress caused by symptoms. This can include fatigue, pain, nausea, and other symptoms.
  Measuring Symptom Burden Symptom Burden Score: (Sum of symptom severity scores / Total number of symptoms assessed) × 100% This can be assessed using symptom scales or questionnaires, where a higher score typically represents a higher symptom burden. Changes in symptom burden are tracked over time to evaluate the effect of the intervention.
Physical Function (6-Minute Walk Test) | From enrollment to the end of treatment at 12 months
  The 6-minute walk test (6MWT) is a measure of a participant's physical endurance and functional capacity, assessing how far they can walk in six minutes. It is often used to evaluate patients with chronic conditions, including those with kidney disease.
  Measuring Physical Function (6-Minute Walk Test) Distance Walked: Total distance walked in six minutes (measured in metres) The result is compared to baseline values or population norms to assess improvements or declines in physical function. A greater distance walked indicates better physical function and endurance.
Cognitive Function (MoCA) | From enrollment to the end of treatment at 12 months
  Cognitive function refers to participants' mental abilities, including memory, attention, reasoning, and problem-solving. This is often measured using cognitive screening tests or detailed neuropsychological assessments.
  Measuring Cognitive Function Cognitive Score: (Sum of individual test scores / Total possible score) × 100% Cognitive function is assessed using tools the Montreal Cognitive Assessment (MoCA). Lower scores may indicate cognitive impairment, while higher scores suggest better cognitive function.
Residual Renal Function (Creatinine Clearance) | From enrollment to the end of treatment at 12 months
  Residual renal function refers to the remaining kidney function in patients who are on dialysis, often measured by creatinine clearance or urine output. Maintaining residual renal function is associated with better outcomes in dialysis patients.
  Measuring Residual Renal Function Residual Renal Function (Creatinine Clearance): Creatinine clearance (measured in mL/min) or urine output (measured in mL/day) Residual renal function is assessed through urine collections or serum creatinine measurements. Higher values suggest better kidney function, and changes are monitored to evaluate the need for adjustments in dialysis.
Restless Legs Syndrome (IRLSSG) | From enrollment to the end of treatment at 12 months
  Restless legs syndrome (RLS) is a neurological condition characterised by an uncontrollable urge to move the legs, often due to uncomfortable sensations. It can significantly impact sleep and quality of life.
  Measuring Restless Legs Syndrome RLS Severity Score: (Sum of individual severity scores from scales like the International Restless Legs Syndrome Study Group (IRLSSG) rating scale / Total possible score) × 100% Higher scores indicate more severe symptoms, and the score is used to monitor the progression or improvement of RLS symptoms over time.
>10g/L Rise in Haemoglobin (Hb) | From enrollment to the end of treatment at 12 months
  This refers to the increase in haemoglobin levels by more than 10g/L over a defined period, typically used as a marker for effective treatment of anemia in conditions like chronic kidney disease or during dialysis.
  Measuring >10g/L Rise in Hb Rise in Hb Rate: (Number of participants with a >10g/L rise in Hb / Total participants enrolled) × 100% This measures the proportion of participants who experience a significant increase in hemoglobin, indicating a positive response to treatment.
% with Haemoglobin >110g/L | From enrollment to the end of treatment at 12 months
  This refers to the proportion of participants who achieve a haemoglobin level greater than 110g/L, often used as a target for managing anaemia in chronic conditions.
  Measuring % with Hb >110g/L Hb >110g/L Rate: (Number of participants with Hb >110g/L / Total participants) × 100% This measure indicates the effectiveness of anaemia management and whether participants are reaching the desired target haemoglobin level.
Ferritin >200ug/L | From enrollment to the end of treatment at 12 months
  Ferritin is a marker of iron stores in the body. A ferritin level greater than 200 ug/L is often used as a target in managing iron levels in patients with chronic kidney disease or anaemia.
  Measuring Ferritin Ferritin Rate: (Number of participants with ferritin >200 ug/L / Total participants) × 100% A higher percentage indicates better iron repletion, while a lower rate suggests suboptimal iron stores, potentially requiring adjustment in treatment.
TSAT >20% | From enrollment to the end of treatment at 12 months
  Transferrin saturation (TSAT) is a measure of iron availability for erythropoiesis. A TSAT greater than 20% is often a target in managing iron deficiency in patients, especially those on dialysis.
  Measuring TSAT TSAT >20 Rate: (Number of participants with TSAT >20% / Total participants) × 100% This rate indicates how many participants are achieving optimal iron saturation, which is crucial for effective anaemia management.
% Receiving Rescue Therapy | From enrollment to the end of treatment at 12 months
  Rescue therapy refers to interventions given to patients who are not responding adequately to the initial treatment. In the context of anaemia management, this might involve additional iron infusions, blood transfusions, or an increase or initiation of erythropoiesis-stimulating agents (ESAs).
  Measuring % Receiving Rescue Therapy Rescue Therapy Rate: (Number of participants receiving rescue therapy / Total participants) × 100% A high rate of participants requiring rescue therapy could indicate that the initial treatment protocol is insufficient or needs adjustment.
Quality-Adjusted Life Years | From enrollment to the end of treatment at 12 months
  Health economics involves evaluating the cost-effectiveness of interventions, considering the economic impact of treatment on the healthcare system, patient quality of life, and outcomes. Data will be collected on additional appointments and admissions.
  Measuring Health Economics Quality-Adjusted Life Years (QALYs): Often used to assess the benefit of a treatment by combining quality of life and survival data.
Change in Erythropoiesis-Stimulating Agent (ESA) Dose | From enrollment to the end of treatment at 12 months
  This refers to the adjustment in the dose of erythropoiesis-stimulating agents (ESA), commonly used to treat anaemia by stimulating red blood cell production in patients with kidney disease.
  Measuring Change in ESA Dose Change in ESA Dose: (Difference in ESA dose before and after treatment) This can be measured as a percentage change from baseline, or as an increase/decrease in units per week. Adjustments are made based on the patient's haemoglobin response.
Cumulative Iron Dose | From enrollment to the end of treatment at 12 months
  The cumulative iron dose refers to the total amount of iron administered over a period, typically used in the treatment of iron deficiency anaemia, especially in patients undergoing dialysis or with chronic kidney disease.
  Measuring Cumulative Iron Dose Cumulative Iron Dose: (Total amount of iron administered over a defined period) This is often tracked in milligrams or grams and can be used to assess the adequacy of iron supplementation and the need for future dosing adjustments. A higher cumulative dose may indicate greater iron deficiency or suboptimal absorption.
Cost per Outcome | From enrollment to the end of treatment at 12 months
  Health economics involves evaluating the cost-effectiveness of interventions, considering the economic impact of treatment on the healthcare system, patient quality of life, and outcomes. Data will be collected on additional appointments and admissions.
  Measuring Health Economics Cost per Outcome: (Total cost of intervention / Total number of successful outcomes) This measure evaluates the economic efficiency of the intervention, with a lower cost per outcome indicating better value for the resources spent.

CONTACTS AND LOCATIONS:
Locations (1):
- Hull University Teaching Hospitals NHS Trust, Hull, East Riding Of Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes